CLINICAL TRIAL: NCT05545488
Title: Examining the Effect of Virtual Reality on Pain and Anxiety Management During Pelvic Examination
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Gülay KURT, Principal Investigator, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2021/20
Record Dates: First submitted 2022-08-22; First posted 2022-09-19 (Actual); Last update posted 2022-09-19 (Actual); Status verified 2022-09

CONDITIONS: Pelvic Examination,Virtual Reality
Keywords: Pelvic Exam; Pain; Anxiety; Virtual Reality
MeSH Terms: conditions — Pain; Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental group (Experimental): Before preparing for pelvic training, information was given about virtual training applications, 1-2 minutes of practical information about both virtual glasses and pelvic training. Afterwards, the woman was taken to the gynecological examination table and, as the doctor began the examination, virtual glasses were put on the woman and a virtual reality application containing both sound and image was performed for 5-15 minutes. In the meantime, the pelvic examination was performed by the physician, the researcher accompanied the woman at all stages of the pelvic examination process and provided care based on ethical principles, which cared for the woman, respected, protected privacy.
  Interventions: Device: Virtual reality
- Control group (No Intervention): The control group was accompanied by the woman at all stages of the pelvic examination process, and the care service that cared for the woman, was respectful, privacy was protected and based on ethical principles was given in the same way, but the virtual glasses initiative was not applied.

INTERVENTIONS:
Device: Virtual reality — I had the women wear virtual reality glasses and watch the video they wanted for at least 5, maximum 15 minutes during the examination.
  Arms: Experimental group

SUMMARY:
Objective: The study was conducted as a randomized controlled experimental study to examine the effect of the video watched with virtual reality glasses during the pelvic examination on the level of pain and anxiety perceived by women.

Materials-Methods: The sample of the study consisted of 128 women (64 experimental, 64 control group) who applied to the Obstetrics and Gynecology Polyclinics with non-pregnancy complaints between November 2021 and February 2022, volunteered to participate in the study and were approved by the doctor for pelvic examination. Institutional and ethical committee permissions were obtained before starting the study. Descriptive Information Form, State Anxiety Scale, Visual Comparison Scale (GDS), Pelvic Examination Experience Evaluation Questionnaire, and Questionnaire Evaluating Non-Verbal Responses to Emotional Stressful Situations, prepared by the researcher, were used to collect data. In the pre-test to the women in the experimental group of the study: Descriptive Information Form, State Anxiety Scale, Visual Comparison Scale (for anxiety), then Pelvic examination + Virtual reality application (using virtual reality glasses for a minimum of 5 maximum 15 minutes), Emotional Stress to be applied by the researcher The Form Evaluating Non-Verbal Responses to the Creating Situations, and in the post-test: State Anxiety Scale, Visual Comparison Scale (anxiety + pain), Pelvic Examination Experience Evaluation Questionnaire were applied. In the pre-test to the women in the control group of the study: Introductory Information Form, State Anxiety Scale, Visual Comparison Scale (for anxiety), then Pelvic examination (routine service), Form Evaluating Non-Verbal Responses to Emotional Stressing Situations to be administered by the Researcher, In the post-test: State Anxiety Scale, Visual Comparison Scale (anxiety + pain), Pelvic Examination Experience Evaluation Questionnaire were applied. Data were evaluated in computer environment and using SPSS 23.0 statistical package program. A p value of <.05 for the data was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18-40
* Being able to read and write
* To be competent to express oneself
* Having applied to the outpatient clinic for any gynecological complaint (bleeding, menstrual cycle irregularity, discharge, itching...) or for routine gynecological control.

Exclusion Criteria:

* Having a current pregnancy
* Complaining of acute pelvic pain
* Having any damage or lesion in the perineum that may cause pain during the examination
* Having used a pharmacological agent or method with analgesic or anxiolytic effect 24 hours before the examination
* Having a vaginismus problem
* Having any physical or mental problems that may prevent communication

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 128 (Actual)
Dates: Start 2021-12-15 (Actual); Primary Completion 2022-02-15 (Actual); Study Completion 2022-03-15 (Actual)

PRIMARY OUTCOMES:
Pain level | 15 minutes
  The visual comparison scale,(VAS).The visual analog scale has a score from 1 to 10. The higher the score, the higher the pain intensity.
Anxiety level | 15 minutes
  The visual comparison scale and the state anxiety scale were evaluated.(VAS).The visual analog scale has a score from 1 to 10. The higher the score, the higher the pain intensity. State Anxiety Scale(STAI FORM TX - I) It is an inventory in which state anxiety is evaluated. The scores vary between 20 and 80 points. With the increase in the score, the level of anxiety also increases.
Pelvic examination using virtual reality glasses | 15 minutes
  Before the video, anxiety is evaluated with a visual comparison scale, then videos with nature, rain, water, flower scenes are watched for 5 to 15 minutes by wearing virtual reality glasses. Afterwards, anxiety and pain are evaluated with state anxiety scale and visual comparison scale. All results SPSS 23.0 It is analyzed by the program.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul University-Cerrahpaşa, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] ACOG Committee Opinion No. 754: The Utility of and Indications for Routine Pelvic Examination. Obstet Gynecol. 2018 Oct;132(4):e174-e180. doi: 10.1097/AOG.0000000000002895. PMID 30247363
- [Background] Bates CK, Carroll N, Potter J. The challenging pelvic examination. J Gen Intern Med. 2011 Jun;26(6):651-7. doi: 10.1007/s11606-010-1610-8. Epub 2011 Jan 12. PMID 21225474
- [Background] Davisson L, Clark K, Powers R, Hobbs G. The rectovaginal examination: physician attitudes and practice patterns. South Med J. 2006 Mar;99(3):212-5. doi: 10.1097/01.smj.0000203334.80885.de. PMID 16553094
- [Background] Granberg S, Wikland M. A comparison between ultrasound and gynecologic examination for detection of enlarged ovaries in a group of women at risk for ovarian carcinoma. J Ultrasound Med. 1988 Feb;7(2):59-64. doi: 10.7863/jum.1988.7.2.59. PMID 3279225
- [Background] Hassan SJ, Sundby J, Husseini A, Bjertness E. The paradox of vaginal examination practice during normal childbirth: Palestinian women's feelings, opinions, knowledge and experiences. Reprod Health. 2012 Aug 28;9:16. doi: 10.1186/1742-4755-9-16. PMID 22929060
- [Background] Ying Lai C, Levy V. Hong Kong Chinese women's experiences of vaginal examinations in labour. Midwifery. 2002 Dec;18(4):296-303. doi: 10.1054/midw.2002.0326. PMID 12473444
- [Background] Mahrer NE, Gold JI. The use of virtual reality for pain control: a review. Curr Pain Headache Rep. 2009 Apr;13(2):100-9. doi: 10.1007/s11916-009-0019-8. PMID 19272275
- [Background] Peeker R, Enerback L, Fall M, Aldenborg F. Recruitment, distribution and phenotypes of mast cells in interstitial cystitis. J Urol. 2000 Mar;163(3):1009-15. PMID 10688040
- [Background] Ueland FR, Depriest PD, Desimone CP, Pavlik EJ, Lele SM, Kryscio RJ, van Nagell JR Jr. The accuracy of examination under anesthesia and transvaginal sonography in evaluating ovarian size. Gynecol Oncol. 2005 Nov;99(2):400-3. doi: 10.1016/j.ygyno.2005.06.030. Epub 2005 Aug 9. PMID 16084576
- [Background] Swahnberg K, Wijma B, Siwe K. Strong discomfort during vaginal examination: why consider a history of abuse? Eur J Obstet Gynecol Reprod Biol. 2011 Aug;157(2):200-5. doi: 10.1016/j.ejogrb.2011.02.025. Epub 2011 Apr 5. PMID 21470763
- [Derived] Kurt G, Ozcan NK. The Effect of Virtual Reality On Pain and Anxiety Management During Pelvic Examination: A Randomized Controlled Trial. J Midwifery Womens Health. 2024 Jul-Aug;69(4):543-549. doi: 10.1111/jmwh.13587. Epub 2024 Jan 4. PMID 38178322